CLINICAL TRIAL: NCT02961608
Title: Conversion Pharmacodynamic Study in Stable Renal Transplant Patients Receiving Tacrolimus Two Times a Day to a New Formulation of Tacrolimus - LCP Tacro - 1 Time a Day.
Acronym: TACPKPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, NURIA LLOBERAS BLANCH, PhD, Hospital Universitari de Bellvitge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACPKPD
Record Dates: First submitted 2016-10-03; First posted 2016-11-11 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Tacrolimus

ARMS (1):
- study group (Experimental)
  Interventions: Drug: Drug conversion from Tacrolimus (Prograf® or Adoport®) to LCP-Tacrolimus (Envarsus®)

INTERVENTIONS:
Drug: Drug conversion from Tacrolimus (Prograf® or Adoport®) to LCP-Tacrolimus (Envarsus®) — Drug conversion from Tacrolimus (Prograf® or Adoport®) to LCP-Tacrolimus (Envarsus®)

SUMMARY:
LCP-Tacro is an extended-release formulation of tacrolimus designed for once-daily dosing. Phase 1 studies demonstrated greater bioavailability than twice-daily tacrolimus capsules and no new safety concerns.

* Stable kidney transplant patients can be safely converted from Adoport® twice-daily to LCP-Tacro®.
* The greater bioavailability of LCP-Tacro after once-daily dosing results in similar (AUC) exposure, at a dose approximately 30% less, than the total daily dose of Adoport®.
* LCP-Tacro provides a slow drug release and this results in flatter kinetics characterized by significantly lower peak-trough fluctuations.
* CN is the major cellular target of the calcineurin inhibitors (CNIs) cyclosporine A (CsA) and tacrolimus. The ability of these drugs to inhibit CN activity is dependent on their binding to the respective immunophilins, cyclophilins A and B for CsA and FKBP12 for tacrolimus.
* CN inhibition is a rate limiting phenomenon. Over concentrations of tacrolimus does not correlate with an increase in the CN activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years).

  * Receivers cadaveric renal graft or living donor with more than 6 months post-transplant evolution.
  * Patients receiving Prograf stable and stable TAC trough concentrations between 5-10ng / ml non-interrupted oral dose for at least 10 days (steady state conditions).
  * receiving concomitant immunosuppressive medication allowed: sodium or mycophenolate mofetil and corticosteroids.
  * Subjects must be willing to give their written informed consent to testing and be able to do consent. If a subject can not give written informed consent independently, you can do your legal representative instead.
  * Women of childbearing age must undergo a pregnancy test at the time of inclusion and accept the use of a medically acceptable method of contraception during the selection and receive medication as specified in the protocol.

Exclusion Criteria:

* • Patients on dialysis or treatment of rejection after transplantation.

  * Patients treated with substances with potential interaction with TAC, particularly potent inhibitors of CYP3A4 (such as telaprevir, boceprevir, ritonavir, ketoconazole, voriconazole, itraconazole, telithromycin or clarithromycin) or inducers of CYP3A4 (such as rifampin or rifabutin).
  * Patients participating in another clinical trial or treated with any investigational drug within 30 days prior to inclusion.
  * Patients with liver disease.
  * The patient or donor with the current diagnosis or history of malignancy within the past 5 years except carcinoma nonmetastatic basal or squamous cell skin treated successfully.
  * pregnant or breast-feeding women and all women of childbearing age unless they use reliable contraception. A pregnancy test will be performed at screening and at the end of the study.
  * Receiver of any other organ transplanted kidney.
  * The recipients of bone marrow or stem cell transplant.
  * Recipients of a kidney from a donor ABO incompatible.
  * Patients with donor specific anti-HLA antibodies.
  * Recipients of a kidney with anticipated cold ischemia time of ≥ 24 hours.
  * Patients with concomitant uncontrolled infection, systemic infection in treatment, or any other unstable medical condition that could interfere with the study objectives.
  * Patients with severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that can affect the absorption of TAC.
  * Patients with white blood cell count ≤ 2.8 x 109 / L unless the absolute neutrophil count (ANC) is ≥ 1.0 x 109 / L
  * Patients with platelet count ≤ 50 x 109 / L
  * Patients with levels of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) exceeding> 3 times the upper limit of normal during the 30 days prior to the transplant procedure.
  * Patients with known hypersensitivity to TAC or any of the excipients in the formulation Envarsus®.
  * unable to swallow study medication patients.
  * Patients with any form of current substance abuse, psychiatric disorder or a condition that, in the investigator's opinion, may invalidate the communication with the investigator.
  * Patients who require a high intake of potassium or potassium-sparing diuretics.
  * Patients treated with substances with known nephrotoxic or neurotoxic effects.
  * positive for hepatitis C virus (HCV-RNA positive) and / or hepatitis B virus (HBV DNA or HBsAg positive) receivers.
  * positive for human immunodeficiency virus (HIV-Ab positive) receivers.
  * unable to understand the effects and risks of the study, who can not give informed consent in writing or unwilling to comply with the study protocol patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of CN activity | Baseline and 35 days post conversion
  The main objective of this study is to compare the area under the curve (AUC) of CN activity after administration of a sustained release formulation (LCP- Tacro, Envarsus®) compared to an immediate release formulation (Prograf®) of TAC in renal transplant patients.

SECONDARY OUTCOMES:
Area Under the curve 0-24 h of each TAC formulation | Baseline and 35 days post conversion
  Pharmacokinetic study AUC 0-24 h of each TAC formulation 12h (Prograf®) and the new formulation of TAC every 24h (LCP- Tacro, Envarsus®).
TAC trough concentrations for optimal inhibition of CN | Baseline and 35 days post conversion
  Study PK / PD: relationship PK TAC (drug exposure) and PD (activity CN) of both formulations. Set TAC trough concentrations for optimal inhibition of CN.
drug exposure according to CYP3A (CYP3A4 and CYP3A5 * 22 * 3) and ABCB1 (C3435T) polymorphism. | Baseline and 35 days post conversion
  Analysis of drug exposure according to CYP3A (CYP3A4 and CYP3A5 * 22 * 3) and ABCB1 (C3435T) polymorphism.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department- Hospital Universitari Bellvtge, L'Hospitalet de Llobregat, Barcelona, Spain